CLINICAL TRIAL: NCT02088723
Title: The Influence of Elevation of the Head of the Bed in Patients With Obstructive Sleep Apnea
Brief Title: Testing the Elevation as Sleep Apnea Treatment
Acronym: TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Apnea-PULMONAR-1
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep
Keywords: Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Polysomnography; Sleep; Patient Positioning
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- head of bed elevation (Experimental): Compare the apnea hypopnea index with the patient in standard polysomnography and in elevated polysomnography (head of bed elevation)
  Interventions: Behavioral: Head of bed elevation

INTERVENTIONS:
Behavioral: Head of bed elevation — head of bed elevation elevation the head of the bed with 15 cm (head of bed elevation) and compare the apnea-hypopnea index with the standard polysomnography

SUMMARY:
The purpose of this study is to determine if the elevation of the head of the bed in patients with obstructive sleep apnea can decrease the apnea-hypopnea index. First the investigators will do a standard polysomnography and see if the patients are included analysing the criteria like apnea-hypopnea index equal or more than 5. Within 2 weeks the patient will do the second polysomnography but this will be with a elevation of the head of the bed (15 cm of elevation of the bed doing a inclination). Then the investigators will compare the data of apnea-hypopnea index in the standard polysomnography versus the index with the elevation of the head of the bed.

DETAILED DESCRIPTION:
There are many researches that demonstrate that the position of the patient modified the apnea-hypopnea index(IAH). In supine position the IAH will increase comparing with lateral position during th sleep. However few studies were done with the elevation of the head of the bed.

First the investigators will do a standard polysomnography and see if the patients are included analysing the criteria like apnea-hypopnea index equal or more than 5. Within 2 weeks the patient will do the second polysomnography but this will be with a elevation of the head of the bed (15 cm of elevation of the bed doing a inclination). Then the investigators will compare the data of apnea-hypopnea index in the standard polysomnography versus the index with the elevation of the head of the bed.The main outcome will be to analyze the apnea hypopnea index comparing standard polysomnography (sPSG) with elevated polysomnography (ePSG).

ELIGIBILITY:
Inclusion Criteria:

* Berlin questionnaire high risk
* Epworth score > 9
* Obstructive Sleep Apnea with an index ≥ 5 events/hour on the polysomnography (The American Academy of Sleep Medicine Manual for the Scoring of Sleep and Associated Events: rules,terminology and technical specifications. American Academy of Sleep Medicine, 2012)

Exclusion Criteria:

* younger than 18 years and older than 80 years
* BMI more than 40 Kg/m2
* heart failure
* renal failure
* uncontrolled respiratory disease
* uncontrolled neurological disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index compared by the polysomnography standard versus polysomnography with the elevation of the head of the bed | The difference between the first exam to the second will be 2 weeks.
  During the polysomnography there are sensors that detect the airflow by cannula pressure and thermistor. WIth those equipment during the all night the patient will be registered and seen if there is absence of flow (apnea) and/or reduction of flow (hypopnea). The apnea and hypopnea index is done by dividing the number of respiratory events by recording time in hours of sleep (events per hour).

CONTACTS AND LOCATIONS:
Overall Officials: Fábio José FB Souza, MD MSc, Principal Investigator — Pulmonar
Locations (1):
- PULMONAR, Criciúma, Santa Catarina, Brazil